CLINICAL TRIAL: NCT05862623
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1 Study of AER-01 (Solution for Inhalation, Delivered Via Nebulizer): As a First-In-Human Single Ascending Dose in Healthy Volunteers (Part A), and a 7-day Multiple Ascending Dose in Healthy Volunteers(Part B)
Brief Title: Single and Multiple Ascending Dose Study of AER-01
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aer Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AER-01-001
Record Dates: First submitted 2023-04-28; First posted 2023-05-17 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2023-08

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AER-01 (Experimental): Specified dose on specified days
  Interventions: Drug: AER-01
- Placebo (Placebo Comparator): Specified dose on specified days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AER-01 — AER-01 solution for inhalation delivered via nebulizer
  Arms: AER-01
Drug: Placebo — Placebo for solution for inhalation delivered via nebulizer
  Arms: Placebo

SUMMARY:
This is a first-in-human, randomized, double-blind, placebo-controlled, Phase 1 study of AER-01 (solution for inhalation, delivered via nebulizer) to assess the safety, tolerability and PK of AER-01. The study will be conducted in 2 parts: a single ascending dose (SAD) part in HVs (Part A) and a 7-day multiple ascending dose (MAD) part in HVs(Part B).

ELIGIBILITY:
Inclusion Criteria Health Volunteers:

* Healthy volunteers: Male or female aged ≥18 to ≤65 years.
* Current non-smoker or casual smoker Participants
* Females must not be pregnant or lactating

Exclusion Criteria:

* History of unstable medical conditions or major surgical procedures over the 12 months prior to Screening.
* History or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic (excluding history of recurrent urinary tract infection), neurologic (excluding history of migraine), dermatologic, psychiatric, renal and/or other major disease or malignancy, or any other condition that in the opinion of the PI or designee might obfuscate the study data.
* History of malignancy of any type, other than in situ cervical cancer or surgically excised non melanomatous skin cancers, within 5 years before Screening. Part B Participants with COPD and Moderate Airflow Limitation
* Has evidence of significant lung restriction on pulmonary function testing or a history of interstitial lung disease (including sarcoidosis and idiopathic pulmonary fibrosis), severe bronchiectasis, cystic fibrosis (asthma is not an exclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Baseline to Day 2 (Part A), Baseline to Day 8 (Part B)
  Will be summarized by cohort, preferred term (PT), system organ class (SOC), severity, and relationship to IP.

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | Baseline to Day 2 (Part A), Baseline to Day 7 (Part B)
  Will be summarized using descriptive statistics by cohort, timepoint, and dose
Time to maximum concentration [Tmax] | Baseline to Day 2 (Part A), Baseline to Day 7 (Part B)
  Will be summarized using descriptive statistics by cohort, timepoint, and dose
Area under the drug concentration-time curve from time 0 (time of dosing) extrapolated to infinity [AUC 0-inf] | Baseline to Day 2 (Part A), Baseline to Day 7 (Part B)
  Will be summarized using descriptive statistics by cohort, timepoint, and dose

CONTACTS AND LOCATIONS:
Overall Officials: Emir Redzepagic, MD, Principal Investigator — CMAX Clinical Research
Locations (2):
- Australia (2):
  - CMAX, Adelaide
  - Scientia Clinical Research, Sydney

IPD SHARING:
Plan to Share IPD: No